CLINICAL TRIAL: NCT06232616
Title: Vitrectomy Combined With Intravitreal Dexamethasone Implant for the Treatment of Idiopathic Epiretinal Membrane With Cystoid Macular Oedema
Brief Title: Vitrectomy Combined With Intravitreal Dexamethasone Implant for Idiopathic Epiretinal Membrane With Macular Oedema
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YFZXYDK202401
Record Dates: First submitted 2024-01-04; First posted 2024-01-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): In this single-arm designed study, participants with idiopathic epiretinal membranes with macular oedema were assigned a vitrectomy with an intravitreal dexamethasone implant.
  Interventions: Procedure: vitrectomy combined with intravitreal dexamethasone implant

INTERVENTIONS:
Procedure: vitrectomy combined with intravitreal dexamethasone implant — The dexamethasone implant will be injected into the vitreous cavity at the end of the surgery.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of 25-gauge pars plana vitrectomy combined with intravitreal dexamethasone implant for the treatment of idiopathic epiretinal membrane with cystoid macular oedema. The main questions it aims to answer are:

* mean changes in best corrected visual acuity and central macular thickness from baseline to post-operative 24 weeks
* mean change in proportion of cystoid macular oedema area from baseline to post-operative 24 weeks
* intraocular pressure throughout postoperative 24 weeks
* concentrations of inflammatory factors in vitreous samples Participants will undergo a standard three-port 25-gauge pars plana vitrectomy and epiretinal membrane peeling combined with phacoemulsification, aspiration, and intraocular lens implantation. The dexamethasone implant will be injected into the vitreous cavity at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients aged 40 years or above with idiopathic stage 3-4 epiretinal membrane defined on the basis of spectral-domain optical coherence tomography classification;
* central retinal thickness >300 µm;
* cystoid oedema within a 1 mm diameter range with the macular fovea as the center;
* ocular axial length less than 25.00 mm.

Exclusion Criteria:

* concomitant or previous macular diseases that may hinder visual improvement other than epiretinal membrane (e.g., age-associated macular degeneration, retinal vein occlusion, or diabetic macular oedema);
* previous vitreoretinal surgery or intravitreal injection history;
* history of glaucoma or optic neuropathy of any kind;
* patients with uncontrolled systemic diseases or infectious diseases;
* patients who took medicines that may have ocular side effects, such as glucocorticoid or hydroxychloroquine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
improvement of visual acuity | from baseline to postoperative 24 weeks
  mean change in best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Ph.D., Study Chair — Shanghai Eye Diseases Prevention & Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
mean change in best corrected visual acuity throughout the study until the results are published in the journal.
Supporting Information: Study Protocol
Time Frame: after the results are published in the journal.
Access Criteria: E-mail contact